CLINICAL TRIAL: NCT07285993
Title: Improving Detection and Outcomes in Patients With Metastatic Invasive Lobular Breast Cancer Through Novel F-18 FAPI PET Imaging
Brief Title: Detection and Outcomes in Metastatic Invasive Lobular Breast Cancer Through Novel F-18 FAP PET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Randy Yeh (Other)
Collaborators: The Society of Nuclear Medicine and Molecular Imaging (Unknown)
Responsible Party: Sponsor-Investigator, Randy Yeh, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-25-00364; PRMC-25-041 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2025-12-11; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Metastatic Invasive Lobular Breast Cancer
Keywords: Breast Cancer; Novel F-18 FAPI PET; Metastatic; Invasive; Lobular; 18F-FDG PET/CT
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FAPI-74 PET/CT and 18F-FDG PET/CT (Experimental): Study participants will undergo both standard-of-care whole body 18F-FDG PET/CT scan and investigational whole-body scan 18F-FAPI-74 PET/CT.
  Interventions: Drug: 18F-FAPI-74; Drug: 18F-FDG; Procedure: PET/CT

INTERVENTIONS:
Drug: 18F-FAPI-74 — FAPI scans will be performed as hybrid PET/CT examinations for attenuation correction and lesion localization. Each patient will be injected intravenously with 7 mCi +/- 2 mCi of 18F-FAPI-74 followed by a 20-minute (+/-10 min) uptake period.
Drug: 18F-FDG — FDG PET/CT will be performed per standard-of-care protocol at Mount Sinai Hospital. Patients will fast for at least 6 hours before FDG administration and plasma glucose levels will be checked to ensure < 200 mg/dL. Each patient will be injected intravenously with 15 mCi +/- 20% of 18F-FDG.
Procedure: PET/CT — FAPI PET/CT images will be acquired from the top of skull to mid-thigh. FDG PET/CT images will be acquired from the skull base to mid-thigh after a 60-min uptake period. Outside FDG PET/CT performed at another institutional can be accepted, if image quality and acquisition is comparable to standard-of-care protocol at Mount Sinai Hospital.

SUMMARY:
This study is a pilot clinical imaging trial of a prospective, head-to-head comparison of 18F-Fibroblast Activation Protein Inhibitor (FAPI)-74 PET/CT versus standard-of-care 18F-Fluorodeoxyglucose (FDG) PET/CT in 15 patients with metastatic invasive lobular breast cancer (ILC). Patients will undergo both 18F-FDG PET/CT and 18F-FAPI-74 PET/CT within a 2-week period (14 days + 7 days) to compare lesions, tumor detection rates, and PET lesion intensity, as well as to assess the clinical value of the PET scans from the treating physician's and the patient's perspective.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Females; Age > 18 years of age
* Diagnosis of invasive lobular breast cancer, with pathologically confirmed metastatic disease.
* ECOG performance status 0-2
* No planned change in anticancer therapy between FDG and FAPI PET scans

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients who cannot undergo PET/CT scanning
* Patients with total serum bilirubin or serum creatinine > 1.5 times the upper limit of normal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of lesions detected by 18F-FAPI-74 PET/CT | End of study, at 1 month
  Proportion of lesions detected by 18F-FAPI-74 PET/CT but not by 18F-FDG PET/CT. All lesions will be mapped across both imaging modalities to determine whether they were detected by FAPI PET/CT but not by FDG PET/CT.

SECONDARY OUTCOMES:
Proportion of lesions detected by 18F-FDG PET/CT but not by 18F-FAPI-74 PET/CT | End of study, at 1 month
  All lesions will be mapped across both imaging modalities to determine whether they were detected by FDG PET/CT but not by FAPI PET/CT.
Proportion of concordant lesions detected by both 18F-FAPI-74 PET/CT and 18F-FDG PET/CT | End of study, at 1 month
  All lesions will be mapped across both imaging modalities to determine whether they were detected by both FAPI PET/CT and FDG PET/CT (i.e., concordant detection).
Tumor detection rate | End of study, at 1 month
  Tumor detection rate, defined as the proportion (%) of patients with >1 lesion on 18F-FAPI-74 PET/CT compared to 18F-FDG PET/CT
SUVmax of the hottest lesion (lesion with highest SUVmax) on 18F-FAPI-74 PET/CT compared to 18F-FDG PET/CT and mean SUVmax across all lesions | End of study, at 1 month
  SUVmax of each lesion identified on both 18F-FAPI-74 PET/CT and 18F-FDG PET/CT.
  Two summary metrics will be derived per patient per modality:
  Hottest lesion SUVmax: Defined as the highest SUVmax value among all detected lesions per patient per modality.
  Overall SUVmax: model lesion-level SUVmax values
Tumor-to-background ratio (TBR) | End of study, at 1 month
  Tumor-to-Background Ratio (TBR) will be defined as the SUVmax of the hottest lesion divided by the SUVmax of two background regions: the liver and the aortic blood pool.
Number of participants with change in therapeutic management decisions | End of study, at 1 month
  Number of participants with change in therapeutic management decisions following review of 18F-FAPI-74 PET/CT compared to decisions based on 18F-FDG PET/CT alone
  For each patient, an initial therapeutic management plan will be recorded based on findings from the 18F-FDG PET/CT scan alone. After the subsequent review of the 18F-FAPI-74 PET/CT scan, a revised management plan will be documented, reflecting any changes informed by the additional imaging data.
Change in disease status assessment | End of study, at 1 month
  Change in disease status assessment (responding, stable, progressing) by treating physicians following review of 18F-FAPI-74 PET/CT compared to assessment based on 18F-FDG PET/CT alone Treating physicians will assign a disease status classification (responding, stable, or progressing) based on available clinical and imaging data from 18F-FDG PET/CT and then after reviewing the 18F-FAPI-74 PET/CT scan. We will summarize the distribution of disease status before and after the FAPI scan, along with the number and percentages of patients whose disease status assessment changed following the FAPI scan, along with the specific nature of those changes.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Yeh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The completed dataset is the sole property of the Sponsor-Investigator's institution and should not be exported to third parties, except for authorized representatives of appropriate Health/Regulatory Authorities, without permission from the Sponsor-investigator and their institution.

REFERENCES:
- [Background] Choi ES, Oh AY, In CB, Ryu JH, Jeon YT, Kim HG. Effects of recruitment manoeuvre on perioperative pulmonary complications in patients undergoing robotic assisted radical prostatectomy: A randomised single-blinded trial. PLoS One. 2017 Sep 6;12(9):e0183311. doi: 10.1371/journal.pone.0183311. eCollection 2017. PMID 28877238
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Fischer S, Dethlefsen S, Klockgether J, Tummler B. Phenotypic and Genomic Comparison of the Two Most Common ExoU-Positive Pseudomonas aeruginosa Clones, PA14 and ST235. mSystems. 2020 Dec 8;5(6):e01007-20. doi: 10.1128/mSystems.01007-20. PMID 33293405
- [Background] Davis AA, Gerratana L, Clifton K, Medford AJ, Velimirovic M, Hensing WL, Bucheit L, Shah AN, D'Amico P, Reduzzi C, Zhang Q, Dai CS, Denault EN, Bagegni NA, Opyrchal M, Ademuyiwa FO, Bose R, Gradishar WJ, Behdad A, Ma CX, Bardia A, Cristofanilli M. Circulating tumour DNA characterisation of invasive lobular carcinoma in patients with metastatic breast cancer. EBioMedicine. 2022 Dec;86:104316. doi: 10.1016/j.ebiom.2022.104316. Epub 2022 Nov 1. PMID 36332363
- [Background] Dumans-Nizard V, Le Guen M, Sage E, Chazot T, Fischler M, Liu N. Thoracic Epidural Analgesia With Levobupivacaine Reduces Remifentanil and Propofol Consumption Evaluated by Closed-Loop Titration Guided by the Bispectral Index: A Double-Blind Placebo-Controlled Study. Anesth Analg. 2017 Aug;125(2):635-642. doi: 10.1213/ANE.0000000000001996. PMID 28537969
- [Background] Benham-Hutchins MM, Effken JA. Multi-professional patterns and methods of communication during patient handoffs. Int J Med Inform. 2010 Apr;79(4):252-67. doi: 10.1016/j.ijmedinf.2009.12.005. Epub 2010 Jan 15. PMID 20079686
- [Background] Niikura N, Costelloe CM, Madewell JE, Hayashi N, Yu TK, Liu J, Palla SL, Tokuda Y, Theriault RL, Hortobagyi GN, Ueno NT. FDG-PET/CT compared with conventional imaging in the detection of distant metastases of primary breast cancer. Oncologist. 2011;16(8):1111-9. doi: 10.1634/theoncologist.2011-0089. Epub 2011 Jul 17. PMID 21765193
- [Background] Dashevsky BZ, Goldman DA, Parsons M, Gonen M, Corben AD, Jochelson MS, Hudis CA, Morrow M, Ulaner GA. Appearance of untreated bone metastases from breast cancer on FDG PET/CT: importance of histologic subtype. Eur J Nucl Med Mol Imaging. 2015 Oct;42(11):1666-1673. doi: 10.1007/s00259-015-3080-z. Epub 2015 May 14. PMID 25971426
- [Background] Hogan MP, Goldman DA, Dashevsky B, Riedl CC, Gonen M, Osborne JR, Jochelson M, Hudis C, Morrow M, Ulaner GA. Comparison of 18F-FDG PET/CT for Systemic Staging of Newly Diagnosed Invasive Lobular Carcinoma Versus Invasive Ductal Carcinoma. J Nucl Med. 2015 Nov;56(11):1674-80. doi: 10.2967/jnumed.115.161455. Epub 2015 Aug 20. PMID 26294295
- [Background] Broudic M, Bodet LM, Dumont R, Joram N, Jacqmarcq O, Caillon J, Flamant C, Thomas C, Tallet A, Piloquet H, Lepelletier D, Gras-Le Guen C, Launay E. A 1-year survey of catheter-related infections in a pediatric university hospital: A prospective study. Arch Pediatr. 2020 Feb;27(2):79-86. doi: 10.1016/j.arcped.2019.11.004. Epub 2019 Nov 29. PMID 31791827
- [Background] Ciriello G, Gatza ML, Beck AH, Wilkerson MD, Rhie SK, Pastore A, Zhang H, McLellan M, Yau C, Kandoth C, Bowlby R, Shen H, Hayat S, Fieldhouse R, Lester SC, Tse GM, Factor RE, Collins LC, Allison KH, Chen YY, Jensen K, Johnson NB, Oesterreich S, Mills GB, Cherniack AD, Robertson G, Benz C, Sander C, Laird PW, Hoadley KA, King TA; TCGA Research Network; Perou CM. Comprehensive Molecular Portraits of Invasive Lobular Breast Cancer. Cell. 2015 Oct 8;163(2):506-19. doi: 10.1016/j.cell.2015.09.033. PMID 26451490
- [Background] Singh M, Jonnalagadda S. Design and characterization of 3D printed, neomycin-eluting poly-L-lactide mats for wound-healing applications. J Mater Sci Mater Med. 2021 Apr 8;32(4):44. doi: 10.1007/s10856-021-06509-7. PMID 33830338
- [Background] Garin-Chesa P, Old LJ, Rettig WJ. Cell surface glycoprotein of reactive stromal fibroblasts as a potential antibody target in human epithelial cancers. Proc Natl Acad Sci U S A. 1990 Sep;87(18):7235-9. doi: 10.1073/pnas.87.18.7235. PMID 2402505
- [Background] Dwyer TJ, Daviskas E, Zainuldin R, Verschuer J, Eberl S, Bye PTP, Alison JA. Effects of exercise and airway clearance (positive expiratory pressure) on mucus clearance in cystic fibrosis: a randomised crossover trial. Eur Respir J. 2019 Apr 18;53(4):1801793. doi: 10.1183/13993003.01793-2018. Print 2019 Apr. PMID 30846472
- [Background] Marchete R, Oliveira S, Bagne L, Silva JIS, Valverde AP, Aro AA, Figueira MM, Fronza M, Bressam TM, Goes VFF, Gaspari de Gaspi FO, Dos Santos GMT, Andrade TAM. Anti-inflammatory and antioxidant properties of Alternanthera brasiliana improve cutaneous wound healing in rats. Inflammopharmacology. 2021 Oct;29(5):1443-1458. doi: 10.1007/s10787-021-00862-3. Epub 2021 Sep 21. PMID 34546478
- [Background] Pase MP, Himali JJ, Mitchell GF, Beiser A, Maillard P, Tsao C, Larson MG, DeCarli C, Vasan RS, Seshadri S. Association of Aortic Stiffness With Cognition and Brain Aging in Young and Middle-Aged Adults: The Framingham Third Generation Cohort Study. Hypertension. 2016 Mar;67(3):513-9. doi: 10.1161/HYPERTENSIONAHA.115.06610. Epub 2016 Jan 11. PMID 26754644
- [Background] Peavy GM, Edland SD, Toole BM, Hansen LA, Galasko DR, Mayo AM. Phenotypic differences based on staging of Alzheimer's neuropathology in autopsy-confirmed dementia with Lewy bodies. Parkinsonism Relat Disord. 2016 Oct;31:72-78. doi: 10.1016/j.parkreldis.2016.07.008. Epub 2016 Jul 21. PMID 27475955
- [Background] Ashworth I, Thielemans L, Chevassut T. Thrombocytopenia: the good, the bad and the ugly. Clin Med (Lond). 2022 May;22(3):214-217. doi: 10.7861/clinmed.2022-0146. PMID 35584828
- [Background] Yokohama T, Iwasaki M, Oura D, Furuya S, Niiya Y. Increased muscle fiber fractional anisotropy value using diffusion tensor imaging after compression without fiber injury. Acta Radiol. 2023 Jan;64(1):139-146. doi: 10.1177/02841851211058282. Epub 2021 Dec 2. PMID 34854736
- [Background] Bremner P, Giuliani M. Impact of resolution, colour, and motion on object identification in digital twins from robot sensor data. Front Robot AI. 2022 Oct 28;9:995342. doi: 10.3389/frobt.2022.995342. eCollection 2022. PMID 36388249
- [Background] [Vasilii Mikhailovich Banshchikov (on his 80th birthday)]. Zh Nevropatol Psikhiatr Im S S Korsakova. 1978;78(5):780-1. No abstract available. Russian. PMID 352072
- [Background] Ishii H, Mukae H, Kadota J, Kaida H, Nagata T, Abe K, Matsukura S, Kohno S. High serum concentrations of surfactant protein A in usual interstitial pneumonia compared with non-specific interstitial pneumonia. Thorax. 2003 Jan;58(1):52-7. doi: 10.1136/thorax.58.1.52. PMID 12511721
- [Background] LHutcheson JA, A Camden, D Charlevoix, T Cushing, M Jochelson, M Kruse, T Langdon, J Levin, C McKay, O Metzger, M Mitchell-Daniels, J Mouabbi, and B Neilsen. . Lobular Breast Cancer Alliance Inc. Survery of Individuals with Metastatatic Invasive Lobular Carcinoma [Poster]. In: Proceedings of the 2022 San Antonio Breast Cancer Symposium.
- [Background] Backhaus P, Gierse F, Burg MC, Buther F, Asmus I, Dorten P, Cufe J, Roll W, Neri D, Cazzamalli S, Millul J, Mock J, Galbiati A, Zana A, Schafers KP, Hermann S, Weckesser M, Tio J, Wagner S, Breyholz HJ, Schafers M. Translational imaging of the fibroblast activation protein (FAP) using the new ligand [68Ga]Ga-OncoFAP-DOTAGA. Eur J Nucl Med Mol Imaging. 2022 May;49(6):1822-1832. doi: 10.1007/s00259-021-05653-0. Epub 2021 Dec 27. PMID 34957527
- [Background] Guyatt GH, Tugwell PX, Feeny DH, Drummond MF, Haynes RB. The role of before-after studies of therapeutic impact in the evaluation of diagnostic technologies. J Chronic Dis. 1986;39(4):295-304. doi: 10.1016/0021-9681(86)90051-2. PMID 3958116